CLINICAL TRIAL: NCT04080687
Title: Effect of Ankle-foot Orthoses on Patients' Confidence in Balance-related Activities
Brief Title: Effect of Ankle-foot Orthoses on Balance Confidence
Acronym: ABCOGS
Status: Completed | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Other Study IDs: URIS201902
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Nerve Disease; Peripheral Nerve Injury Lower Limb; Poliomyelitis; Cerebral Palsy; Multiple Sclerosis
Keywords: ankle-foot orthoses; lower limbs; rehabilitation outpatients; balance confidence; falls
MeSH Terms: conditions — Peripheral Nervous System Diseases; Poliomyelitis; Cerebral Palsy; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers: The patients who had fallen during the 6 months prior to the study onset
  Interventions: Device: Ankle-foot orthosis
- Non-fallers: The patients who had not fallen during the 6 months prior to the study onset
  Interventions: Device: Ankle-foot orthosis

INTERVENTIONS:
Device: Ankle-foot orthosis — Ankle-foot orthosis of any type (unilateral or bilateral, standard or carbon fiber, for support or correction)

SUMMARY:
The patients at our Prosthetics and Orthotics Outpatient Clinic who have had an ankle-foot orthosis for at least one year will fill in the Activities-Specific Balance Confidence Scale (ABC Scale) for wearing the orthosis and for not wearing the orthosis. They will also answer a mini survey about falls in order to determine whether they have fallen within the last 6 months.

DETAILED DESCRIPTION:
The effect of the orthosis will be estimated as the difference between the two ABC Scale scores. The ABC Scale score and individual items will be compared between the fallers and the non-fallers.

ELIGIBILITY:
Inclusion Criteria:

* patients at our Prosthetics and Orthotics Outpatient Clinic having an ankle-foot orthosis for at least 1 year

Exclusion Criteria:

* insufficient cognitive ability to fill in the ABC Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients of our Prosthetics and Orthotics Outpatient Clinic who have had an ankle-foot orthosis for at least 1 year and able to fill in the ABC Scale
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
ABC Scale | At day 0
  Activities-Specific Balance Confidence Scale (ABC Scale) will be filled in for the confidence without the orthosis and confidence with the orthosis. The ABC Scale is a 16-item self-report measure in which patients rate their balance confidence for performing activities. Each item is rated on a scale from 0 (no confidence) to 100 (complete confidence). Overall score is the average rating across the items.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Burger, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No